CLINICAL TRIAL: NCT03880812
Title: Does Societal Cost Information Affect Patient Decision-Making in Carpal Tunnel Syndrome: A Randomized Controlled Trial
Brief Title: Cost Information on Carpal Tunnel Syndrome Treatment Decisions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: Stanford University (Other)
Responsible Party: Principal Investigator, David Ring, Associate Dean for Comprehensive Care and Professor, Department of Surgery and Perioperative Care, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-09-0067
Record Dates: First submitted 2019-03-13; First posted 2019-03-19 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Intervention Model Description: Patients were randomized in an intervention group that reviewed societal costs associated with carpal tunnel release and a control group that did not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cost group (Experimental): These patients reviewed total societal costs associated with carpal tunnel release.
  Interventions: Other: Societal cost
- No cost group (No Intervention): These patients did not review total societal costs associated with carpal tunnel release.

INTERVENTIONS:
Other: Societal cost — Annual societal cost information to the US for carpal tunnel release surgery was displayed.
  Arms: Cost group

SUMMARY:
The purpose of this study was to determine whether the provision of societal cost information affects patients' decisions whether or not to undergo surgical management in carpal tunnel syndrome, using a hypothetical scenario.

DETAILED DESCRIPTION:
Given the large societal costs of carpal tunnel surgery and existence of a relatively inexpensive treatment option, carpal tunnel release provides fertile ground for testing whether societal costs can influence patient decision-making in hand surgery. Such work would inform future efforts to reduce societal healthcare costs by elucidating whether appeals to societal cost are effective at driving stewardship of limited healthcare resources at the patient level. In this study, the investigators aimed to answer this question by presenting participants with a hypothetical scenario in which the participants had to choose between surgery and wrist bracing for carpal tunnel syndrome. Participants were randomized into two cohorts and societal cost information was presented to the intervention group. The effect of societal cost information on treatment choice is assessed, along with participants' healthcare attitudes.

ELIGIBILITY:
Inclusion Criteria:

* English speaking upper extremity patients
* Nontraumatic condition

Exclusion Criteria:

* Traumatic condition

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2018-09-24 (Actual); Primary Completion 2018-12-26 (Actual); Study Completion 2018-12-26 (Actual)

PRIMARY OUTCOMES:
Number of participants choosing carpal tunnel release or splinting | Immediately after reading the hypothetical scenario
  Choice for carpal tunnel release over splinting. All participants were presented a hypothetical case of mild carpal tunnel syndrome. The scenario described (nocturnal) symptoms of numbness and tingling and two treatment choices: carpal tunnel release or wrist splinting. In addition, participants were randomized to review total annual societal cost information for CTR procedures in the United States. After reviewing the case, participants were asked to indicate if they would choose surgery (more expensive) or splinting (less expensive). Scoring was measured on a 6-point ordinal Likert scale (ranging from 1="Definitely not" to 6="Definitely").

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Austin Regional Clinic, Austin, Texas
  - Texas Orthopedics, Austin, Texas
  - HTB Musculoskeletal Institute, Austin, Texas
  - Seton Institute for Plastic and Reconstructive Surgery, Austin, Texas
  - Orthopedic Specialists of Austin, Austin, Texas
  - ATX Ortho, Austin, Texas

IPD SHARING:
Plan to Share IPD: No